CLINICAL TRIAL: NCT05647785
Title: Extension Study to Compare Long-term Efficacy of Two Digital Software Medical Devices as Interventions for Physical and Mental Health in Cancer Patients Previously Enrolled in the RESTORE Study
Brief Title: Long-term Follow-up of RESTORE Study
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Blue Note Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT005
Record Dates: First submitted 2022-11-28; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- cerena™: Subjects who took part in the cerena™ group during the original RESTORE study
  Interventions: Device: Long-term follow-up of cerena™
- attune™: Subjects who took part in the attune™ group during the original RESTORE study
  Interventions: Device: Long-term follow-up of attune™

INTERVENTIONS:
Device: Long-term follow-up of cerena™ — Long term follow-up for eligible participants from the RESTORE study
  Groups: cerena™
Device: Long-term follow-up of attune™ — Long term follow-up for eligible participants from the RESTORE study
  Groups: attune™

SUMMARY:
The RESTORE extension study is a non-interventional, long-term follow-up study with people who participated in the study referred to as RESTORE (NCT05227898).

The purpose of this extension study is to understand the durability of the effects of two digital software devices on anxiety and other indicators of psychological and physical health in participants of the RESTORE study in the 6-months after study completion.

Subjects who were enrolled and not withdrawn from the original RESTORE study are eligible to participate. People who consent to participate will be asked to electronically complete a set of questionnaires at 3 months and 6 months following the scheduled date of their RESTORE end-of-study visit.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in and not withdrawn from the original RESTORE study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of all interested patients who were enrolled and not withdrawn from the parent study (RESTORE).
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2022-10-31 (Actual); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Symptoms of anxiety | 3 and 6 months post RESTORE end-of-study
  The PROMIS-Anxiety (PROMIS-A) is a validated PRO consisting of 8 questions measuring anxiety symptoms. The change in PROMIS-A score over time will be assessed (reduction indicates reduced anxiety).

SECONDARY OUTCOMES:
Symptoms of depression | 3 and 6 months post RESTORE end-of-study
  The PROMIS-Depression (PROMIS-D) is a validated PRO consisting of 8 questions measuring depression symptoms. The change in PROMIS-D score over time will be assessed (decrease indicates reduced depression).
Symptoms of emotional distress | 3 and 6 months post RESTORE end-of-study
  Change in PROMIS Emotional Distress; a composite of PROMIS-Anxiety and PROMIS-Depression over time (decrease indicates reduced emotional distress).
Cancer-related symptoms of anxiety (intrusions) | 3 and 6 months post RESTORE end-of-study
  The Impact of Events Scale-Revised (IES-R) is used to assess subjective distress caused by a stressful life event, which in this study is cancer. The change in the IES-R Intrusion subscale score over time will be assessed (decrease indicates reduced intrusive symptoms related to cancer).
Wellbeing and quality of life | 3 and 6 months post RESTORE end-of-study
  The Functional Assessment of Cancer Therapy - General (FACT-G) is designed to measure four domains of HRQOL in cancer patients: Physical, social, emotional, and functional well-being. The change in FACT-G scores over time will be assessed (increase indicates improved quality of life).
Stress management/coping skills | 3 and 6 months post RESTORE end-of-study
  The Measure of Current Status (MOCS) Part A measures self-perceived status for using coping skills. The change in MOCS Part A scores over time will be assessed (increase indicates greater confidence in skill use ability).
Non-specific (social) intervention effects | 3 and 6 months post RESTORE end-of-study
  The Measure of Current Status (MOCS) Part B assesses non-specific intervention effects - feelings of normalcy vs. alienation, sense of cohesiveness with other patients, perceptions of care from persons around them, and a sense of being better off than other cancer patients. The change in MOCS Part B scores over time will be assessed (increase indicates greater non-specific intervention effects).
Perceived stress | 3 and 6 months post RESTORE end-of-study
  The Perceived Stress Scale (PSS) measures how different situations affect feelings and perceived stress. The change in PSS scores over time will be assessed (higher PSS scores indicate higher perceived stress).
Benefit finding | 3 and 6 months post RESTORE end-of-study
  The 17-item Benefit Finding Scale measures the perception that positive contributions were made to one's life by the experience of being diagnosed with and treated for cancer. Change in scores over time will be assessed (increase indicates increase in benefit finding).

OTHER OUTCOMES:
Fear of cancer recurrence | 3 and 6 months post RESTORE end-of-study
  The Fear of Cancer Recurrence Inventory - Short Form and the Fear of Cancer Recurrence single item measure assess the fear of cancer returning or progressing (higher scores indicate greater fear of cancer recurrence).
Healthcare utilization - visits and admissions | 3 and 6 months post RESTORE end-of-study
  Number of visits and admissions (higher indicates greater healthcare utilization)
Healthcare utilization - hospitalizations | 3 and 6 months post RESTORE end-of-study
  Length of hospitalizations in days (higher indicates greater healthcare utilization)
Healthcare utilization - medications | 3 and 6 months post RESTORE end-of-study
  Number of medications (higher indicates greater healthcare utilization)
Healthcare utilization - claims and costs | 3 and 6 months post RESTORE end-of-study
  Number of healthcare claims and associated costs (higher indicates greater healthcare utilization)

CONTACTS AND LOCATIONS:
Overall Officials: Dianne M Shumay, PhD, Principal Investigator — Blue Note Therapeutics
Locations (1):
- Blue Note Therapeutics, San Francisco, California, United States